CLINICAL TRIAL: NCT04098003
Title: INvestigation of the Gut microbiomE and STatin Response (INGEST)
Brief Title: Investigation of the Gut Microbiome and Statin Response
Acronym: INGEST
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sony Tuteja (Other)
Responsible Party: Sponsor-Investigator, Sony Tuteja, Research Assistant Professor of Medicine, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 832874
Record Dates: First submitted 2019-09-13; First posted 2019-09-20 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers
Keywords: gut microbiome; statins; cholesterol
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This is a randomized, placebo controlled, double blind (participant and outcomes assessor) trial to investigate the effects of rosuvastatin on the gut microbiome. Healthy volunteers will be randomized to rosuvastatin 20 mg daily or placebo for eight weeks in a 2:1 ratio.
Who Masked: Participant, Outcomes Assessor
Masking Description: Matching placebo capsules will be formulated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rosuvastatin (Experimental): rosuvastatin 20 mg daily for eight weeks
  Interventions: Drug: Rosuvastatin
- Placebo (Placebo Comparator): placebo daily for eight weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — rosuvastatin 20 mg daily or placebo for eight weeks
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — Matched placebo control
  Arms: Placebo

SUMMARY:
There is evidence that the bacteria that naturally reside in the gut can influence how well we respond to medications. Therefore this study will look at how rosuvastatin, a medication used to lower cholesterol levels, may change the bacteria in the gut. Investigators will also examine how the gut bacteria will affect the ability of rosuvastatin to lower cholesterol levels. There will be 4 study visits over the course of about 16 weeks.The expected duration of the study is 2 years. Investigators plan to enroll 100 healthy volunteers during that time.

DETAILED DESCRIPTION:
The gut microbiome plays an important role in the metabolism of xenobiotics and contributes to the variation in drug response. Atorvastatin, simvastatin and rosuvastatin, three of the most commonly prescribed statin medications, also display evidence for modulation by the gut microbiome.The objective of this study is to understand the interaction between the gut microbiome and host drug response to statin therapy using 16S rRNA sequencing, metagenomics sequencing and bile acid metabolomics.

Aim 1: To compare changes in the gut microbiome in healthy volunteers randomized to an 8-week intervention with rosuvastatin 10mg daily or placebo.

Aim 2: To determine the relationship with gut microbiome, fecal bile acid composition, serum FGF19 levels and the change in plasma LDL-C with rosuvastatin.

This is a randomized, placebo controlled trial to investigate the effects of rosuvastatin on the gut microbiome, fecal bile acids and FGF19 levels. Healthy volunteers will be randomized to rosuvastatin 20 mg daily or placebo for eight weeks in a 2:1 ratio. Participants will be blinded to treatment assignment. Stool and blood will be collected at baseline, 8 weeks, and 12 weeks for 16S sequencing, plasma lipid assays, bile acid metabolites and FGF19 assays. A subgroup of participants at the tails of LDL-C response will undergo metagenomics sequencing.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is capable of giving informed consent
2. Participant is aged 18 to 65 years. The gut microbiome has been shown to change gradually with time, although there is no cut-off in age when this occurs.

Exclusion Criteria:

1. Participants with cardiovascular disease such as a history of heart failure (New York Heart Association class II-IV), myocardial infarction, stroke, coronary artery bypass graft, hypertension, and hyperlipidemia as these conditions are associated with altered gut microbiome composition.74 Hypertension is defined as blood pressure greater than 160/110 or on any anti-hypertensive medications. LDL-C >190 mg/dl or <100 mg/dl and triglycerides > 400 mg/dl.
2. Participants with a history of cancer.
3. Kidney disease (serum creatinine >1.5 mg/dl).
4. Liver dysfunction (alanine aminotransferase > 2 times the upper limit of normal).
5. Diabetes mellitus (DM) - Diabetes itself may affect the gut microbiome although this has not been extensively studied. In addition to a prior diagnosis of diabetes mellitus other than that related to pregnancy, a fasting glucose level of greater than 125mg/dL will be used to exclude participation.
6. Clinical diagnosis of hypothyroidism
7. History of inflammatory disorders of the intestinal tract (i.e. IBD, celiac sprue).
8. Use of antibiotics in the prior 6 months.
9. Use of pre-, pro-, or synbiotics.
10. Chronic medication use (including over the counter medications and herbal supplements) with the exception of oral contraceptives. Since we are evaluating the impact of rosuvastatin on the gut microbiome we would like to exclude the potential impact of confounding medications.
11. Current smoker. The effect of smoking on the microbiome of the gut is unknown.
12. Known history of alcohol or substance abuse.
13. Body Mass Index (BMI) <18.5 or >30 kg/m2. Volunteers with BMI below normal will be excluded to prevent inclusion of subjects with a subclinical systemic disease that may influence the gut microbiome. Volunteers with moderate or severe obesity will be excluded as obesity may be associated with altered gut microbiome composition.31
14. Unable to abstain from consumption of illicit drugs during the study period.
15. Prior bowel resection surgery other than appendectomy. It is unknown how prior bowel resection surgery may influence the microbiome composition; hence we will exclude these participants.
16. Baseline bowel frequency less than every 2 days or greater than 3 times daily. Normal bowel frequency is every 3rd day to 3 times per day. Although unknown, stool frequency could be related to the microbiome composition. To avoid the need for use of antidiarrheal medications or laxatives, which themselves could alter the microbiome composition, these patients will be excluded.
17. Participant has experienced diarrhea within the two weeks prior to entry. Diarrhea is defined as a change in bowel habits with an increased frequency or loose stools such that the stool could not be lifted with a fork.
18. Vegans and Vegetarians.
19. Known intolerance to statin medications.
20. Unwilling to obtain from grapefruit containing foods or drinks.
21. Pregnant women. To avoid any risk to an unborn fetus from study drug exposure.
22. Refusal to use two medically accepted method of birth control while participating in the study, such as a barrier method, hormonal contraceptives, implanted birth control devices, permanent methods (such as a vasectomy), and/or abstinence.
23. Nursing mothers
24. Any condition that the investigator feels may limit the volunteer's ability to complete the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in bacterial abundance | 8 weeks
  as measured by operational taxonomic units (OTUs)

SECONDARY OUTCOMES:
Change in LDL-C | 8 weeks
  low density lipoprotein cholesterol levels (mg/dl)

OTHER OUTCOMES:
Change in fecal bile acid concentrations | 8 weeks
  concentration of bile acids (nM)
Change in serum FGF19 levels | 8 weeks
  Fibroblast growth factor 19 levels (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Sony Tuteja, PharmD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Phildelphia, Pennsylvania, United States